CLINICAL TRIAL: NCT03981822
Title: A Phase 2, Double-Blind, Placebo-Controlled Study to Determine the Dose Regimen, Efficacy, Safety, and Tolerability of VP-102 in Subjects With External Genital Warts
Brief Title: A Placebo-Controlled Study Using VP-102 in the Treatment of External Genital Warts
Acronym: CARE-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verrica Pharmaceuticals Inc. (Industry)
Collaborators: Instat Consulting, Inc. (Other); Paidion Research, Inc. (Industry); BioClinica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-102-104
Record Dates: First submitted 2019-06-06; First posted 2019-06-11 (Actual); Results first posted 2021-09-22 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2021-08

CONDITIONS: Condylomata Acuminata; Papillomavirus Infections; Skin Diseases, Viral; Skin Diseases, Infectious; Skin Diseases; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases; Warts
Keywords: Human Papilloma Virus (HPV); Genital Warts; Sexually Transmitted Disease (STD); Viral Disease
MeSH Terms: conditions — Condylomata Acuminata; Papillomavirus Infections; Skin Diseases, Viral; Skin Diseases, Infectious; Skin Diseases; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases; Warts; Virus Diseases | interventions — VP-102; Cantharidin

STUDY DESIGN:
Intervention Model Description: The aim of Part A is to determine the two best treatment regimens for evaluation of safety and efficacy in Part B. Increasing durations of skin exposure to study drug (VP-102 or placebo) will be evaluated in three treatment groups (n=6/group) that will enroll progressively.
  Part B of the study will begin enrollment only after the Sponsor has selected the two dose regimens in Part A, which will be called VP-102 Regimen 1 and Regimen 2.Approximately 90 subjects will be enrolled and randomized to one of four treatment arms (two treatment regimens, each with VP-102 and Placebo). Randomization will be stratified by sex so that neither gender exceeds ~60% of any treatment arm. Two of the treatment arms will be VP-102 Regimen 1 and VP-102 Regimen 2. The other two treatment arms will be placebo (Placebo Regimen 1 and Placebo Regimen 2), with corresponding durations of skin exposure matching those selected for VP-102 Regimen 1 and Regimen 2.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (8):
- Part A: VP-102 2 hour-Active (Active Comparator): For part A, VP-102 will be applied for 2 hours and removed. If selected as a dose regimen for Part B VP-102 will be applied for 2 hours and removed.In both parts, VP-102 is applied every 21 days for 4 treatments.
  Interventions: Combination Product: VP-102 and applicator
- Part A: VP-102 6-hour Active (Active Comparator): For part A, VP-102 will be applied for 6 hours and removed. If selected as a dose regimen for Part B VP-102 will be applied for 6 hours and removed. In both parts, VP-102 is applied every 21 days for 4 treatments.
  Interventions: Combination Product: VP-102 and applicator
- Part A: VP-102 24-hour Active (Active Comparator): For part A, VP-102 will be applied for 24 hours and removed. If selected as a dose regimen for Part B, VP-102 will be applied for 24 hours and removed. In both parts, VP-102 is applied every 21 days for 4 treatments.
  Interventions: Combination Product: VP-102 and applicator
- Part A: Placebo (Placebo Comparator): For part A, VP-102 will be applied for 2-,6- or 24- hours and removed. Placebo is applied every 21 days for 4 treatments.
  Interventions: Combination Product: Placebo
- Part B & A: VP-102 6 hour-Active (Active Comparator): Part B, VP-102 will be applied for 6 hours and removed. VP-102 is applied every 21 days for 4 treatments.
  Interventions: Combination Product: VP-102 and applicator
- Part B & A: 6-hour-Placebo (Placebo Comparator): Part B, Placebo will be applied for 6 hours and removed. VP-102 is applied every 21 days for 4 treatments.
  Interventions: Combination Product: Placebo
- Part B & A: VP-102 24-hour Active (Active Comparator): For part A, VP-102 will be applied for 24 hours and removed. If 24 hours is selected as a dose regimen for Part B, VP-102 will be applied for 24 hours and removed. VP-102 is applied every 21 days for 4 treatments.
  Interventions: Combination Product: VP-102 and applicator
- Part B & A: 24-hour-Placebo (Placebo Comparator): Part B, VP-Placebo will be applied for 24 hours and removed. VP-102 is applied every 21 days for 4 treatments.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: VP-102 and applicator — In part A, VP-102 will be applied for either 2, 6 or 24 hours with each regimen compared to placebo. For part B, 2 of the regimens from part A will be chosen for Part B with each compared to Placebo. Only 4 arms are actually being studied.
  Other Names: VP-102 (cantharidin) 0.7% w/v topical solution
  Arms: Part A: VP-102 2 hour-Active; Part A: VP-102 24-hour Active; Part A: VP-102 6-hour Active; Part B & A: VP-102 24-hour Active; Part B & A: VP-102 6 hour-Active
Combination Product: Placebo — The placebo single-use applicator contains the same formulation as the VP-102 applicator but does not contain the active pharmaceutical ingredient cantharidin
  Arms: Part A: Placebo; Part B & A: 24-hour-Placebo; Part B & A: 6-hour-Placebo

SUMMARY:
This is a Phase 2, double-blind, placebo-controlled study to determine the dose regimen, safety, tolerability, and efficacy of VP-102 in subjects with External Genital Warts (EGW). This study is divided into two parts (Part A and Part B). Increasing durations of skin exposure to study drug (VP-102 or placebo) will be evaluated in three treatment groups prior to progressing to enrollment in Part B. Part A & B will enroll a approximately 108 subjects completing 4 treatment applications every 21 days and continuing with follow-up assessments at Day 84, 112 and 147.

DETAILED DESCRIPTION:
This study is to determine the Dose Regimen, Efficacy, Safety, and Tolerability of VP-102 in Subjects with External Genital Warts. It is divided into two parts (Part A and Part B). The aim of Part A is to determine the two best treatment regimens for evaluation of safety and efficacy in Part B.In Part A, Study drug (VP-102 or placebo) will be administered once every 21 days for up to four applications. Enrollment will begin in Group 1, then proceed into Group 2, and lastly into Group 3. A safety review will be conducted to determine whether enrollment can be initiated into the next Group. An additional blinded safety review will be performed after all six subjects in Group 3 have completed the 48-hour Visit, in order to support dose selection for Part B (Safety and Efficacy). Part B of the study will begin enrollment only after the Sponsor has selected the two dose regimens from Part A. The study will remain blinded until completion of both parts of the study.

In Part A, up to 18 subjects will be randomized to VP-102 or placebo treatment with three different regimens. When Part B is open an additional ~90 subjects will be enrolled and randomized to VP-102 or placebo with two treatment regimens. Two of the treatment arms will be VP-102 Regimen 1 and VP-102 Regimen 2. The other two treatment arms will be placebo (Placebo Regimen 1 and Placebo Regimen 2), with corresponding durations of skin exposure matching those selected for VP-102 Regimen 1 and Regimen 2. As an example, if the regimens selected from Part A are the 2-hour and 6-hour applications of VP-102, then VP-102 Regimen 1 would be VP-102 treatment for 2-hours and VP-102 Regimen 2 would be VP-102 treatment for 6-hours. Likewise, Placebo Regimen 1 would be placebo treatment for 2 hours and Placebo Regimen 2 would be placebo treatment for 6-hours. Randomization of the four treatment arms (VP-102 Regimen 1:VP-102 Regimen 2:Placebo Regimen 1:Placebo Regimen 2) will be 3:3:2:2. In both Regimen 1 and Regimen 2, study drug will be administered to EGW once every 21 days for up to four applications. Subjects will be asked to remove the study drug at the designated time selected from the dose regimen findings in Part A of the study. Treatment will continue with a minimum of every 21 days, until complete clearance or a maximum of four treatment sessions. Safety assessments including recording of local skin reactions are conducted at each treatment visit and at follow up visits Day 84, 112, and 147.

ELIGIBILITY:
Key Inclusion Criteria:

* Be healthy, immunocompetent males or females ≥ 18 years of age
* Present with ≥ 2 and ≤ 30 external genital and/or perianal warts in ≥ 1 of the following anatomic areas:

  * In both sexes: medial thigh (except inguinal fold); supra-pubic, perineal, and perianal areas
  * In men: over the glans penis (excluding urethral meatus), penis shaft, scrotum, and foreskin
  * In women: vulva (excluding labia minora and mucosal surfaces)
* Have warts present for ≥ 4 weeks at the baseline visit
* Have warts that are ≤ 8 mm in diameter each

Key Exclusion Criteria:

* Have a wart within the allowed treatment area > 8 mm in diameter or with an eroded or ulcerated surface, in the Investigator's opinion
* Have an unclear diagnosis of condyloma
* Have any wart types other than genital warts (e.g., common or plantar warts) that require treatment during the study period
* Have active genital herpes eruption, or had active genital herpes lesions within 4 weeks before enrollment
* Have a history of neoplasia or other HPV-associated malignancies within the last 5 years
* Are systemically immunosuppressed
* Are sexually active or may become sexually active and are unwilling to practice responsible birth control methods
* Are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Guenthner, MD, Principal Investigator — The Indiana Clinical Trials Center
Locations (4):
- United States (4):
  - The Indiana Clinical Trials Center,PC, Plainfield, Indiana
  - DelRicht Research, Baton Rouge, Louisiana
  - Clarkston Skin Research, Clarkston, Michigan
  - DelRicht Research, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guenthner S, McFalda W, Tate M, Eads K, Rieger J, Glover DK, Willson C, Rumney P, Rosen T, Andres J, Olivadoti M. Phase II, Double-Blind, Vehicle-Controlled Study to Determine the Cantharidin Dose Regimen, Efficacy, Safety, and Tolerability of VP-102 in Subjects with External Genital Warts. Am J Clin Dermatol. 2021 Nov;22(6):867-875. doi: 10.1007/s40257-021-00635-2. Epub 2021 Sep 13. PMID 34515985

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 groups from Part A were to be included in Part B based on Part A analysis.
Pre-assignment Details: All subject numbers are based on ITT population. Participants in Part A 6-hour and 24-hour group were also included in Part B subject populations.
Groups:
- Part A: VP-102 2-hour; Part A: VP-102 6-hour Group; Part A: VP-102 24-hour Group: VP-102 and applicator: In part A, VP-102 will be applied for either 2, 6 or 24 hours with each regimen compared to placebo. For part B, 2 of the regimens from part A will be chosen for Part B with each compared to Placebo. Only 4 arms are actually being studied.
- Part A: Placebo: This includes 3 subjects that received placebo (1 each for the 2-hour; 6-hour and 24-hour)
- Part B: VP-102 6-hour; Part B: VP-102 24-hour: VP-102 and applicator: For part B, 2 of the regimens from part A will be chosen for Part B with each compared to Placebo. Only 4 arms are actually being studied.
- Part B: Placebo 6-hour; Part B: Placebo 24-hour: Placebo and applicator: For part B, 2 of the regimens from part A will be chosen for Part B with each compared to Placebo. Only 4 arms are actually being studied.
Period: Overall Study
Arm/Group | Part A: VP-102 2-hour | Part A: VP-102 6-hour Group | Part A: VP-102 24-hour Group | Part A: Placebo | Part B: VP-102 6-hour | Part B: Placebo 6-hour | Part B: VP-102 24-hour | Part B: Placebo 24-hour
Started | 5 | 5 | 5 | 3 | 25 | 23 | 22 | 17
Completed | 5 | 3 | 4 | 3 | 17 | 17 | 16 | 12
Not Completed | 0 | 2 | 1 | 0 | 8 | 6 | 6 | 5
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 6 | 4 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — COVID-19 Related | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Part A: VP-102 2-hour: VP-102 will be applied for 2-hours and removed. VP-102 is applied every 21 days for 4 treatments.
- Part A: VP-102 6-hour; Part B: VP-102 6-hour: VP-102 will be applied for 6-hours and removed. VP-102 is applied every 21 days for 4 treatments.
- Part A: VP-102 24-hour; Part B: VP-102 24-hour: VP-102 will be applied for 24-hours and removed. VP-102 is applied every 21 days for 4 treatments.
- Part A: Placebo: Placebo will be applied for 2-,6- or 12-hours and removed. Placebo is applied every 21 days for 4 treatments.
- Part B: 6-hour-Placebo: Placebo will be applied for 6-hours and removed. VP-102 is applied every 21 days for 4 treatments.
- Part B: 24-hour-Placebo: Placebo will be applied for 24-hours and removed. VP-102 is applied every 21 days for 4 treatments.
- Total: Total of all reporting groups
Arm/Group | Part A: VP-102 2-hour | Part A: VP-102 6-hour | Part A: VP-102 24-hour | Part A: Placebo | Part B: VP-102 6-hour | Part B: 6-hour-Placebo | Part B: VP-102 24-hour | Part B: 24-hour-Placebo | Total
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 25 | 23 | 22 | 17 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.40 (9.915) | 43.00 (8.246) | 33.80 (5.263) | 32.00 (3.606) | 38.12 (10.138) | 35.87 (7.973) | 34.45 (7.526) | 33.88 (6.470) | 35.85 (8.260)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 0 | 10 | 10 | 10 | 7 | 46
  Male | 1 | 2 | 3 | 3 | 15 | 13 | 12 | 10 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 6 | 1 | 2 | 5 | 15
  Not Hispanic or Latino | 4 | 5 | 5 | 3 | 19 | 22 | 20 | 12 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 0 | 6 | 8 | 1 | 6 | 24
  White | 3 | 5 | 3 | 3 | 19 | 12 | 21 | 11 | 77
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 3 | 25 | 23 | 22 | 17 | 105
Baseline number of treatable external genital warts [Mean (Standard Deviation); unit: genital warts] | 7 (5.568) | 9.60 (12.012) | 13.00 (8.276) | 11.67 (12.423) | 8.28 (6.380) | 5.87 (3.684) | 8.68 (5.489) | 7.76 (6.897) | 8.08 (6.395)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Exhibiting Complete Clearance of All Treatable Warts at the Study Day 84 (End of Treatment) Visit.
Description: Proportion of subjects exhibiting complete clearance of all treatable warts (baseline and new) at the Study Day 84 EOT Visit.
Time Frame: Compares baseline wart count to Day 84, end of treatment.
Population: Part B and A: Intent-to-Treat Population. Part B summary is pooled with its respective treatments from Part A.
Measure: Count of Participants; unit: Participants
Groups:
- Part B Pooled With Part A: VP-102 6-hour; Part B Pooled With Part A: Placebo 6-hour; Part B Pooled With Part A VP-102 24-hour; Part B Pooled With Part A: Placebo 24-hour: Data will be summarized for both Part B pooled with Part A for the applicable treatments.
Arm/Group | Part B Pooled With Part A: VP-102 6-hour | Part B Pooled With Part A: Placebo 6-hour | Part B Pooled With Part A VP-102 24-hour | Part B Pooled With Part A: Placebo 24-hour
Number analyzed (Participants) | 30 | 24 | 27 | 18
Participants
  Yes | 11 | 1 | 9 | 0
  No | 19 | 23 | 18 | 18
Statistical Analysis 1: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0048, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 2: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0075, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender

2. Secondary Outcome: Proportion of Subjects Exhibiting Complete Clearance of All Treatable Warts (Baseline and New) at Treatment Visit 2, Treatment Visit 3, Treatment Visit 4, and Follow-up Visits on Study Day 112 and Study Day 147 (EOS)
Description: Proportion of subjects exhibiting complete clearance of all treatable warts (baseline and new) at Treatment Visit 2, Treatment Visit 3, Treatment Visit 4, and Follow-up Visits on Study Day 112 and Study Day 147 (EOS).
Time Frame: Clearance compared from baseline to each study visit, treatment 2 (Day 21), 3 (Day 42), 4 (Day 63) and Day 84, 112 and 147.
Population: Part B and A pooled - ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Pooled With Part A: VP-102 6-hour | Part B Pooled With Part A: Placebo 6-hour | Part B Pooled With Part A VP-102 24-hour | Part B Pooled With Part A: Placebo 24-hour
Number analyzed (Participants) | 30 | 24 | 27 | 18
Participants
  Treatment Visit 2: Yes, Complete Clearance | 1 | 0 | 4 | 0
  Treatment Visit 3: Yes, Complete Clearance | 4 | 0 | 8 | 2
  Treatment Visit 4: Yes, Complete Clearance | 6 | 0 | 7 | 0
  Study Day 84 EOT: Yes, Complete Clearance | 11 | 1 | 9 | 0
  F/U Visit Day 112: Yes, Complete Clearance | 9 | 2 | 8 | 2
  F/U Visit Day 147: Yes, Complete Clearance | 6 | 3 | 8 | 2
Statistical Analysis 1: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 2 - Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.3642, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 2: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 2: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0967, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 3: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 3: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0648, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 4: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 3: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.1357, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 5: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 4 Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0190, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender. Part B summary is pooled with its respective treatments from
Statistical Analysis 6: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 4 Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0184, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 7: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Study Day 84 EOT Visit - Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0048, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 8: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Study Day 84 EOT Visit - Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0075, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 9: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Follow-up Visit Day 112 - Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0539, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 10: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow-up Visit Day 112 - Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.1638, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 11: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Follow-up Visit Day 147 EOS - Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.4766, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 12: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow-up Visit Day 147 EOS - Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.1588, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender

3. Secondary Outcome: Proportion of Subjects Exhibiting 90% Clearance of All Treatable Warts (Baseline and New) at Treatment Visit 2, Treatment Visit 3, Treatment Visit 4, Study Day 84 (EOT), and Follow-up Visits on Study Day 112 and Study Day 147 (EOS)
Description: Proportion of subjects exhibiting 90% clearance of all treatable warts (baseline and new) at Treatment Visit 2, Treatment Visit 3, Treatment Visit 4, Study Day 84 (EOT), and Follow-up Visits on Study Day 112 and Study Day 147 (EOS).
Time Frame: Compared from baseline to each study visit, treatment 2 (Day 21), 3 (Day 42), 4 (Day 63) and Day 84, 112 and 147.
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Pooled With Part A: VP-102 6-hour | Part B Pooled With Part A: Placebo 6-hour | Part B Pooled With Part A VP-102 24-hour | Part B Pooled With Part A: Placebo 24-hour
Number analyzed (Participants) | 30 | 24 | 27 | 18
Participants
  Treatment Visit 2: Incidence of >=90% Clearance: YES | 1 | 0 | 4 | 0
  Treatment Visit 3: Incidence of >=90% Clearance: YES | 5 | 0 | 8 | 2
  Treatment Visit 4: Incidence of >=90% Clearance: YES | 7 | 0 | 7 | 0
  Study Day 84 EOT: Incidence of >=90% Clearance: YES | 14 | 2 | 11 | 0
  F/U Visit Day 112: Incidence of >=90% Clearance: YES | 11 | 2 | 9 | 2
  F/U Visit Day 147: Incidence of >=90% Clearance: YES | 9 | 3 | 9 | 2
Statistical Analysis 1: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 2 Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.3642, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender. Part B summary is pooled with its respective treatments from Part A
Statistical Analysis 2: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 3 Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0356, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 3: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 4 Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0118, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 4: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Study Day84 EOT Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0026, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 5: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Follow-up Visit Day 112 Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0174, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 6: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Follow-up Visit Day 147 EOS Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.1311, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 7: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 2 Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0967, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 8: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 3 Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.1357, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 9: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 4 Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0184, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 10: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Study Day 84 EOT Visit Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0024, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 11: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow-up Visit Day 112 Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.1034, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 12: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow-up Visit Day 147 EOS Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.1029, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender

4. Secondary Outcome: Proportion of Subjects Exhibiting 75% Clearance of All Treatable Warts (Baseline and New) at Treatment Visit 2, Treatment Visit 3, Treatment Visit 4, Study Day 84 (EOT), and Follow-up Visits on Study Day 112 and Study Day 147 (EOS)
Description: Proportion of subjects exhibiting 75% clearance of all treatable warts (baseline and new) at Treatment Visit 2, Treatment Visit 3, Treatment Visit 4, Study Day 84 (EOT), and Follow-up Visits on Study Day 112 and Study Day 147 (EOS).
Time Frame: Compared from baseline to each study visit, treatment 2, (Day 21), 3 (Day 42), 4 (Day 63) and Day 84, 112 and 147.
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Pooled With Part A: VP-102 6-hour | Part B Pooled With Part A: Placebo 6-hour | Part B Pooled With Part A VP-102 24-hour | Part B Pooled With Part A: Placebo 24-hour
Number analyzed (Participants) | 30 | 24 | 27 | 18
Participants
  Treatment Visit 2: Incidence of >=75% Clearance: YES | 5 | 0 | 6 | 1
  Treatment Visit 3: Incidence of >=75% Clearance: YES | 8 | 0 | 14 | 2
  Treatment Visit 4: Incidence of >=75% Clearance: YES | 11 | 2 | 12 | 1
  Study Day 84 EOT: Incidence of >=75% Clearance: YES | 15 | 2 | 15 | 2
  F/U Visit Day 112: Incidence of >=75% Clearance: YES | 13 | 3 | 13 | 3
  F/U Visit Day 147: Incidence of >=75% Clearance: YES | 10 | 4 | 13 | 2
Statistical Analysis 1: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 2: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0356, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 2: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 2: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.1477, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 3: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 3: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0062, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 4: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 3: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0046, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 5: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 4: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0177, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 6: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 4: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0054, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 7: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Study Day 84 (EOT) visit: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 8: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Study Day 84 (EOT) Visit: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0034, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 9: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Follow-up visit day 112: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0156, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 10: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow-up visit day 112: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0367, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 11: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Follow-up visit day 147 (EOS): Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.1746, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender
Statistical Analysis 12: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow-up visit day 147 (EOS): Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0123, Cochran-Mantel-Haenszel; P-value is based on the CMH test stratified by gender

5. Secondary Outcome: Change From Baseline in the Number of Treatable Warts (Baseline and New) at Treatment Visit 2, Treatment Visit 3, Treatment Visit 4, Study Day 84 (EOT), and Follow-up Visits on Study Day 112 and Study Day 147 (EOS)
Description: Change from baseline in the number of treatable warts (baseline and new) at Treatment Visit 2, Treatment Visit 3, Treatment Visit 4, Study Day 84 (EOT), and Follow-up Visits on Study Day 112 and Study Day 147 (EOS).
  Number of warts present were recorded at each treatment visit as well as follow-up visits. For each post baseline treatment visit, the change in number of warts from baseline was calculated.
Time Frame: Compared from baseline to each study visit, treatment 2 (Day 21), 3 (Day 42), 4 (Day 63) and Day 84, 112 and 147.
Population: ITT Populations
Measure: Mean (Standard Deviation); unit: Warts
Arm/Group | Part B Pooled With Part A: VP-102 6-hour | Part B Pooled With Part A: Placebo 6-hour | Part B Pooled With Part A VP-102 24-hour | Part B Pooled With Part A: Placebo 24-hour
Number analyzed (Participants) | 30 | 24 | 27 | 18
Warts
  Treatment Visit 2: number analyzed (Participants) | 28 | 23 | 23 | 18
  Treatment Visit 2 | -4.0 (4.95) | -0.3 (1.11) | -5.3 (4.25) | 0.6 (30.07)
  Treatment Visit 3: number analyzed (Participants) | 25 | 23 | 23 | 15
  Treatment Visit 3 | -4.4 (5.80) | -1.1 (3.69) | -6.3 (5.45) | -0.5 (5.01)
  Treatment Visit 4: number analyzed (Participants) | 25 | 23 | 18 | 13
  Treatment Visit 4 | -5.2 (4.72) | -0.9 (3.98) | -7.1 (5.09) | 0.5 (5.17)
  Study Day 84 EOT Visit: number analyzed (Participants) | 21 | 21 | 20 | 13
  Study Day 84 EOT Visit | -6.1 (5.24) | -1.1 (4.92) | -7.4 (6.37) | 0.1 (5.12)
  Follow up Day 112: number analyzed (Participants) | 21 | 19 | 19 | 14
  Follow up Day 112 | -5.3 (5.21) | -1.1 (5.33) | -8.1 (5.54) | -0.3 (4.39)
  Follow-up Visit Day 147 EOS: number analyzed (Participants) | 17 | 17 | 20 | 12
  Follow-up Visit Day 147 EOS | -5.0 (7.63) | -1.2 (5.49) | -7.9 (5.46) | -0.1 (4.66)
Statistical Analysis 1: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 2: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0021, Mixed Models Analysis — Analysis is based on MMRM model; MMRM model with gender, Tx, visit, Tx by visit interaction, and baseline wart count as factors. An unstructured covariance model was used; LS mean difference = -3.96, 95% CI 2-sided [-5.41 to -1.24]
Statistical Analysis 2: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 3: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0150, Mixed Models Analysis; MMRM model with gender, Tx, visit, treatment by visit interaction, and baseline wart count as factors. An unstructured covariance model was used; LS mean difference = -4.72, 95% CI 2-sided [-5.95 to -0.66]
Statistical Analysis 3: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 4: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0011, Mixed Models Analysis — Analysis is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -5.31, 95% CI 2-sided [-6.54 to -1.69]
Statistical Analysis 4: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Study Day 84 EOT Visit: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0007, Mixed Models Analysis — P-value is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -6.50, 95% CI 2-sided [-8.25 to -2.32]
Statistical Analysis 5: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Follow-up day 112: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0012, Mixed Models Analysis — P-value is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -6.15, 95% CI 2-sided [-7.50 to -1.91]
Statistical Analysis 6: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Follow-up visit day 147 (EOS): Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0349, Mixed Models Analysis — P-value is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -5.02, 95% CI 2-sided [-6.78 to -0.26]
Statistical Analysis 7: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment visit 2: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p < 0.0001, Mixed Models Analysis — P-value is based on MMRM mode; [statistical method as in outcome 5, analysis 2]; LS mean difference = -4.76, 95% CI 2-sided [-7.47 to -2.85]
Statistical Analysis 8: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 3: Degrees of freedom associated with the error term were computed using Kenward-Rogers method; Test type: Superiority; p = 0.0005, Mixed Models Analysis — Analysis is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -6.00, 95% CI 2-sided [-8.37 to -2.43]
Statistical Analysis 9: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment visit 4: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Analysis based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -6.64, 95% CI 2-sided [-9.65 to -4.12]
Statistical Analysis 10: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Study Day 84 (EOT): Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0004, Mixed Models Analysis — Analysis is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -6.49, 95% CI 2-sided [-9.67 to -2.92]
Statistical Analysis 11: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow-up day 112: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Analysis based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -6.96, 95% CI 2-sided [-9.89 to -3.57]
Statistical Analysis 12: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow up day 147 (EOS): Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0005, Mixed Models Analysis — Analysis based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -6.99, 95% CI 2-sided [-10.20 to -2.94]

6. Secondary Outcome: Percent Change From Baseline in the Number of Treatable Warts (Baseline and New) at Treatment Visit 2, Treatment Visit 3, Treatment Visit 4, at Study Day 84 (EOT), and Follow-up Visits on Study Day 112 and Study Day 147 (EOS)
Description: Percent Change from Baseline in the Number of Treatable Warts (Baseline and New) at Treatment Visit 2, Treatment Visit 3, Treatment Visit 4, at Study Day 84 (EOT), and Follow-up Visits on Study Day 112 and Study Day 147 (EOS).
Time Frame: Percent change from baseline to each study visit, treatment 2 (Day 21), 3 (Day 42), 4 (Day 63) and Day 84, 112 and 147.
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Wart percentage change from Baseline
Arm/Group | Part B Pooled With Part A: VP-102 6-hour | Part B Pooled With Part A: Placebo 6-hour | Part B Pooled With Part A VP-102 24-hour | Part B Pooled With Part A: Placebo 24-hour
Number analyzed (Participants) | 30 | 24 | 27 | 18
Wart percentage change from Baseline
  Treatment Visit 2: number analyzed (Participants) | 28 | 23 | 23 | 18
  Treatment Visit 2 | -41.4 (32.38) | -6.2 (13.14) | -58.5 (26.69) | -2.6 (30.07)
  Treatment Visit 3: number analyzed (Participants) | 25 | 23 | 23 | 15
  Treatment Visit 3 | -49.0 (37.18) | -8.9 (44.46) | -69.3 (34.03) | -17.8 (49.79)
  Treatment Visit 4: number analyzed (Participants) | 25 | 23 | 18 | 13
  Treatment Visit 4 | -65.8 (30.69) | -5.1 (66.26) | -77.3 (26.87) | 0.6 (41.94)
  Study Day 84 End of Treatment Visit: number analyzed (Participants) | 21 | 21 | 20 | 13
  Study Day 84 End of Treatment Visit | -79.7 (34.27) | -1.6 (78.34) | -77.1 (38.66) | -5.5 (47.98)
  Follow up Day 112: number analyzed (Participants) | 21 | 19 | 19 | 14
  Follow up Day 112 | -68.2 (43.20) | 1.9 (91.11) | -79.2 (28.36) | -14.2 (49.60)
  Follow up Visit Day 147 End of Study: number analyzed (Participants) | 17 | 17 | 20 | 12
  Follow up Visit Day 147 End of Study | -42.5 (111.83) | -6.0 (86.56) | -79.6 (25.01) | -12.9 (50.49)
Statistical Analysis 1: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 2: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p < 0.0001, Mixed Models Analysis — P-value is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -41.47, 95% CI 2-sided [-51.31 to -20.87]
Statistical Analysis 2: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 3: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0004, Mixed Models Analysis — P-value is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -50.95, 95% CI 2-sided [-66.18 to -19.56]
Statistical Analysis 3: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 4: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p < 0.0001, Mixed Models Analysis — P-value is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -66.21, 95% CI 2-sided [-88.15 to -35.87]
Statistical Analysis 4: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Study Day 84 End of Treatment Visit: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p < 0.0001, Mixed Models Analysis — P-value is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -79.37, 95% CI 2-sided [-111.44 to -49.77]
Statistical Analysis 5: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Follow up Day 112: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0001, Mixed Models Analysis — P-value is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -69.79, 95% CI 2-sided [-103.17 to -35.25]
Statistical Analysis 6: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Follow up Visit Day 147 End of Study: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.1033, Mixed Models Analysis — P-value is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -41.22, 95% CI 2-sided [-90.61 to 8.56]
Statistical Analysis 7: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 2: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p < 0.0001, Mixed Models Analysis — P-value is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -58.43, 95% CI 2-sided [-73.26 to -39.39]
Statistical Analysis 8: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 3: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p < 0.0001, Mixed Models Analysis — P-value is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -69.86, 95% CI 2-sided [-81.61 to -28.80]
Statistical Analysis 9: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 4: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p < 0.0001, Mixed Models Analysis — P-value is based on MMRM model with gender, treatment, visit, treatment by visit interaction, and baseline wart count as factors; [statistical method as in outcome 5, analysis 2]; LS mean difference = -76.55, 95% CI 2-sided [-107.19 to -45.61]
Statistical Analysis 10: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Study Day 84 End of Treatment Visit: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0003, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 9]; [statistical method as in outcome 5, analysis 2]; LS mean difference = -74.29, 95% CI 2-sided [-102.96 to -31.55]
Statistical Analysis 11: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow-up Day 112: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0004, Mixed Models Analysis — P-value is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -77.10, 95% CI 2-sided [-110.32 to -32.78]
Statistical Analysis 12: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow-up Visit Day 147 End of Study: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0178, Mixed Models Analysis — P-value is based on MMRM model; [statistical method as in outcome 5, analysis 2]; LS mean difference = -77.52, 95% CI 2-sided [-120.82 to -11.88]

7. Other Pre Specified Outcome: Proportion of Subjects Exhibiting Reduction of ≥ 1 Treatable Wart From Baseline at Treatment Visit 2, Treatment Visit 3, Treatment Visit 4, Study Day 84 (EOT), and Follow-up Visits on Study Day 112 and Study Day 147 (EOS)
Description: Proportion of subjects exhibiting reduction of ≥ 1 treatable wart from baseline at Treatment Visit 2, Treatment Visit 3, Treatment Visit 4, Study Day 84 (EOT), and Follow-up Visits on Study Day 112 and Study Day 147 (EOS).
Time Frame: Compared from baseline to each study visit, treatment 2 (Day 21), 3 (Day 42), 4 (Day 63) and Day 84, 112 and 147.
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Pooled With Part A: VP-102 6-hour | Part B Pooled With Part A: Placebo 6-hour | Part B Pooled With Part A VP-102 24-hour | Part B Pooled With Part A: Placebo 24-hour
Number analyzed (Participants) | 30 | 24 | 27 | 18
Participants
  Treatment Visit 2: Yes - at least 1 wart reduction from Baseline | 22 | 6 | 23 | 6
  Treatment Visit 2: No | 8 | 18 | 4 | 12
  Treatment Visit 3: Yes - at least 1 wart reduction from Baseline | 20 | 10 | 21 | 7
  Treatment Visit 3: No | 10 | 14 | 6 | 11
  Treatment Visit 4: Yes - at least 1 wart reduction from Baseline | 23 | 10 | 17 | 4
  Treatment Visit 4: No | 7 | 14 | 10 | 14
  Study Day 84 EOT Visit: Yes - at least 1 wart reduction from Baseline | 19 | 9 | 18 | 4
  Study Day 84 EOT Visit: No | 11 | 15 | 9 | 14
  F/U Visit Day 112: Yes - at least 1 wart reduction from Baseline | 17 | 10 | 18 | 5
  F/U Visit Day 112: No | 13 | 14 | 9 | 13
  F/U Visit Day 147 EOS: Yes - at least 1 wart reduction from Baseline | 13 | 8 | 19 | 5
  F/U Visit Day 147 EOS: No | 17 | 16 | 8 | 13
Statistical Analysis 1: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 2: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 2: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 2: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 3: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 3: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0698, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 4: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 3: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0100, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 5: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Treatment Visit 4: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0101, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 6: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Treatment Visit 4: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0077, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 7: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Study Day 84 EOT Visit: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0640, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 8: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Study Day 84 EOT: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0045, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 9: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Follow-up Visit Day 112: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.2840, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 10: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow-up Visit Day 112: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0132, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 11: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Follow-up Visit Day 147 EOS: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.4668, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender
Statistical Analysis 12: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow-up Visit Day 147 EOS: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0064, Cochran-Mantel-Haenszel — P-value is based on the CMH test stratified by gender

8. Other Pre Specified Outcome: Proportion of Subjects Who Are Clear at the Study Day 84 (End of Treatment) Visit and Remain Clear at the Follow-up Visits on Study Day 112 and Study Day 147 (End of Study)
Description: Proportion of subjects who are clear at all three study visits, Study Day 84 (End of Treatment) Visit and remain clear at the Follow-up Visits on Study Day 112 and Study Day 147 (End of Study).
Time Frame: Complete clearance compared from Day 84 to follow-up days 112 and 147.
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Pooled With Part A: VP-102 6-hour | Part B Pooled With Part A: Placebo 6-hour | Part B Pooled With Part A VP-102 24-hour | Part B Pooled With Part A: Placebo 24-hour
Number analyzed (Participants) | 30 | 24 | 27 | 18
Participants
  Yes | 5 | 0 | 7 | 0
  No | 25 | 24 | 20 | 18
Statistical Analysis 1: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0364, Mantel Haenszel; Stratified by gender
Statistical Analysis 2: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0215, Cochran-Mantel-Haenszel; Stratified by gender

9. Other Pre Specified Outcome: Change From Baseline in Total Wart Area (Sum of Individual Warts) at Study Day 84 (EOT), and Follow-up Visits on Study Day 112 and Study Day 147 (EOS)
Description: Change from baseline in total wart area (sum of individual warts) at Study Day 84 (EOT), and Follow-up Visits on Study Day 112 and Study Day 147 (EOS).
Time Frame: Baseline to Study Day 84, Follow-up Visits at Days 112 and 147 (EOS)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Part B Pooled With Part A: VP-102 6-hour | Part B Pooled With Part A: Placebo 6-hour | Part B Pooled With Part A VP-102 24-hour | Part B Pooled With Part A: Placebo 24-hour
Number analyzed (Participants) | 30 | 24 | 27 | 18
mm^2
  Study Day 84 (EOT): number analyzed (Participants) | 10 | 20 | 11 | 13
  Study Day 84 (EOT) | -52.60 (67.067) | -23.64 (59.722) | -72.87 (91.659) | 1.60 (33.796)
  Follow-up Day 112: number analyzed (Participants) | 12 | 17 | 11 | 12
  Follow-up Day 112 | -79.43 (99.679) | -20.35 (53.289) | -82.79 (71.750) | 1.40 (39.963)
  Follow-up Visit Day 147 (EOS): number analyzed (Participants) | 11 | 14 | 12 | 10
  Follow-up Visit Day 147 (EOS) | -59.28 (100.988) | -6.02 (36.929) | -68.78 (68.710) | 2.21 (45.035)
Statistical Analysis 1: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Study Day 84 (EOT: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.1222, Mixed Models Analysis — Analysis is based on MMRM model; MMRM model with gender, Tx, visit, treatment by visit interaction, and baseline wart area as factors. An unstructured covariance model was used; LS mean difference = -59.63, 95% CI 2-sided [-76.10 to 9.23]
Statistical Analysis 2: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Study Day 112 (EOT: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0403, Mixed Models Analysis — Analysis based on MMRM model; [statistical method as in outcome 9, analysis 1]; LS mean difference = -69.51, 95% CI 2-sided [-81.30 to -1.90]
Statistical Analysis 3: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Follow-up Visit Day 147 (EOS): Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0863, Mixed Models Analysis — Analysis is based on MMRM model; [statistical method as in outcome 9, analysis 1]; LS mean difference = -58.88, 95% CI 2-sided [-77.79 to 5.33]
Statistical Analysis 4: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Study Day 84 (EOT): Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0428, Mixed Models Analysis — Analysis is based on MMRM model; [statistical method as in outcome 9, analysis 1]; LS mean difference = -62.13, 95% CI 2-sided [-100.76 to -1.73]
Statistical Analysis 5: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow-up Day 112: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0084, Mixed Models Analysis — Analysis is based on MMRM model; [statistical method as in outcome 9, analysis 1]; LS mean difference = -71.93, 95% CI 2-sided [-110.46 to -17.00]
Statistical Analysis 6: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow-up Visit Day 147 (EOS): Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0273, Mixed Models Analysis — Analysis is based on MMRM model; [statistical method as in outcome 9, analysis 1]; LS mean difference = -63.11, 95% CI 2-sided [-103.08 to -6.35]

10. Other Pre Specified Outcome: Percent Change From Baseline in the Total Wart Area (Sum of Individual Warts) at Study Day 84 (EOT), and Follow-up Visits on Study Day 112 and Study Day 147 (EOS)
Description: Percent Change from baseline in the total wart area (sum of individual warts) at Study Day 84 (EOT), and Follow-up Visits on Study Day 112 and Study Day 147 (EOS).
Time Frame: Baseline to Study Day 84 (EOT), and Follow-up Visits on Study Day 112 and Study Day 147 (EOS)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Change from baseline in % of wart area
Arm/Group | Part B Pooled With Part A: VP-102 6-hour | Part B Pooled With Part A: Placebo 6-hour | Part B Pooled With Part A VP-102 24-hour | Part B Pooled With Part A: Placebo 24-hour
Number analyzed (Participants) | 30 | 24 | 27 | 18
Change from baseline in % of wart area
  Study Day 84 (EOT): number analyzed (Participants) | 10 | 20 | 11 | 13
  Study Day 84 (EOT) | -46.0 (52.77) | -22.3 (57.92) | -64.2 (55.78) | -7.3 (93.42)
  Follow-up Day 112: number analyzed (Participants) | 12 | 17 | 11 | 12
  Follow-up Day 112 | -48.2 (54.67) | -21.5 (64.54) | -76.4 (12.33) | 13.8 (129.61)
  Follow-up Day 147 (EOS): number analyzed (Participants) | 11 | 14 | 12 | 10
  Follow-up Day 147 (EOS) | -45.8 (71.37) | -11.7 (52.52) | -69.3 (16.44) | 19.9 (138.49)
Statistical Analysis 1: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Study Day 84 (EOT): Part B summary is pooled with its respective treatments from Part A; Test type: Superiority — Analysis is based on MMRM model; p = 0.3083, Mixed Models Analysis; [statistical method as in outcome 9, analysis 1]; LS mean difference = -44.65, 95% CI 2-sided [-69.96 to 22.47]
Statistical Analysis 2: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Follow-up Day 112: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.1686, Mixed Models Analysis — Analysis is based on MMRM model; [statistical method as in outcome 9, analysis 1]; LS mean difference = -55.80, 95% CI 2-sided [-86.93 to 15.56]
Statistical Analysis 3: Comparison: Part B Pooled With Part A: VP-102 6-hour vs Part B Pooled With Part A: Placebo 6-hour; Follow-up Visit Day 147 End of Study: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.2384, Mixed Models Analysis — Analysis is based on MMRM model; [statistical method as in outcome 9, analysis 1]; LS mean difference = -38.06, 95% CI 2-sided [-87.04 to 22.10]
Statistical Analysis 4: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Study Day 84 (EOT): Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0603, Mixed Models Analysis — Analysis is based on MMRM model; [statistical method as in outcome 9, analysis 1]; LS mean difference = -61.96, 95% CI 2-sided [-103.37 to 2.27]
Statistical Analysis 5: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow-up Visit Day 112: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0109, Mixed Models Analysis — Analysis is based on MMRM model; [statistical method as in outcome 9, analysis 1]; LS mean difference = -74.87, 95% CI 2-sided [-138.71 to -18.83]
Statistical Analysis 6: Comparison: Part B Pooled With Part A VP-102 24-hour vs Part B Pooled With Part A: Placebo 24-hour; Follow-up Visit Day 147 End of Study: Part B summary is pooled with its respective treatments from Part A; Test type: Superiority; p = 0.0467, Mixed Models Analysis — Analysis is base on MMRM model; [statistical method as in outcome 9, analysis 1]; LS mean difference = -66.62, 95% CI 2-sided [-127.64 to -0.99]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected following the first application of study drug through Study Day 147.
Description: TEAEs defined as those AEs that occurred after dosing and those existing AEs that worsened during the study. Subject numbers in the AE summaries differ from the participant flow module based on the differences in the ITT population and the safety population. Due to randomization system errors, one subject was randomized to VP-102 6-hour but received VP-102 24-hour. Two subjects were randomized to Placebo 6-hour but received Placebo 24-hour.
Groups:
- Part A: VP-102 2-hour; Part A: Placebo 2-hour: Data summarized for VP-102 2-hour group.
Arm/Group | Part B Pooled With Part A: VP-102 6-hour | Part B Pooled With Part A: Placebo 6-hour | Part B Pooled With Part A VP-102 24-hour | Part B Pooled With Part A: Placebo 24-hour | Part A: VP-102 2-hour | Part A: Placebo 2-hour
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/22 | 0/28 | 0/20 | 0/5 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/22 | 0/28 | 1/20 | 0/5 | 0/1
Other Adverse Events (participants affected / at risk) | 29/29 | 15/22 | 28/28 | 9/20 | 5/5 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part B Pooled With Part A: VP-102 6-hour (N=29) | Part B Pooled With Part A: Placebo 6-hour (N=22) | Part B Pooled With Part A VP-102 24-hour (N=28) | Part B Pooled With Part A: Placebo 24-hour (N=20) | Part A: VP-102 2-hour (N=5) | Part A: Placebo 2-hour (N=1)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part B Pooled With Part A: VP-102 6-hour (N=29) | Part B Pooled With Part A: Placebo 6-hour (N=22) | Part B Pooled With Part A VP-102 24-hour (N=28) | Part B Pooled With Part A: Placebo 24-hour (N=20) | Part A: VP-102 2-hour (N=5) | Part A: Placebo 2-hour (N=1)
Application site vesicles (General disorders) | 25 | 0 | 26 | 1 | 4 | 0
Application site pain (General disorders) | 20 | 3 | 19 | 4 | 4 | 0
Application site erythema (General disorders) | 14 | 3 | 19 | 1 | 2 | 0
Application site pruritus (General disorders) | 14 | 5 | 10 | 1 | 1 | 0
Application site scab (General disorders) | 13 | 1 | 14 | 0 | 1 | 0
Application site discolouration (General disorders) | 7 | 4 | 6 | 0 | 4 | 0
Application site dryness (General disorders) | 7 | 2 | 6 | 1 | 1 | 0
Application site erosion (General disorders) | 6 | 0 | 7 | 0 | 4 | 0
Application site oedema (General disorders) | 3 | 1 | 7 | 1 | 3 | 0
Application site exfoliation (General disorders) | 3 | 2 | 5 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Major Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Umbilical hernia repair (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Due to logistical and/or scheduling difficulties related to the SARS-CoV-2 (coronavirus-19; COVID-19) pandemic during the course of the study, six subjects discontinued due to COVID-19 related reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is bound to terms and conditions of a Sponsored Clinical Trial Agreement which has strict confidentiality obligations running to Sponsor and broad provisions restricting PI's rights to publish or present any data or Study Results without Sponsor's express review consent and review.

DOCUMENTS (2):
  • Study Protocol (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT03981822/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT03981822/SAP_001.pdf